CLINICAL TRIAL: NCT06203951
Title: Improving Perinatal Outcomes Among Kenyan Pregnant Women With an Integrated STI Testing Model
Acronym: PrIMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jillian Pintye, Associate Professor, Department of Biobehavioral Nursing and Health Informatics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00019163; R01HD113455-01A1 (NIH)
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hiv; Sexually Transmitted Infections (Not HIV or Hepatitis)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (No Intervention): In all arms, participants will receive syndromic STI assessment from study nurses at the antenatal clinic per Kenyan national guidelines, which entails a clinician (i.e., nurse, physician, clinical officer) using an algorithm asking whether clients have symptoms of vaginal discharge, lower abdominal pain, or genital ulcers followed by a physical examination for signs that match the self-reported symptoms. Based on clinical presentation, treatment is prescribed. Study nurses will capture information on symptoms, treatment acceptance, and dispensation. All participants will be provided with a study phone number to call at any time free of charge for clarifying questions or concerns with STI medication use.
- Universal Testing (Experimental): Participants randomized to universal STI testing will be offered Xpert® CT/NG and TV testing regardless of symptoms, and they will receive a standard syndromic STI assessment.
  Interventions: Diagnostic Test: Xpert® CT/NG and TV testing
- Asymptomatic Only Testing (Experimental): Participants randomized to the asymptomatic only testing will be offered Xpert® CT/NG and TV testing if no signs or symptoms of CT, NG, or TV are identified during STI assessment.
  Interventions: Diagnostic Test: Xpert® CT/NG and TV testing

INTERVENTIONS:
Diagnostic Test: Xpert® CT/NG and TV testing — Participants randomized to universal STI testing will be offered Xpert® CT/NG and TV testing regardless of symptoms, and they will receive a standard syndromic STI assessment. Participants randomized to the asymptomatic only testing will be offered Xpert® CT/NG and TV testing if no signs or symptoms of CT, NG, or TV are identified during STI assessment. Participants assigned to receive Xpert® testing will be counseled on CT/NG/TV testing, including the benefits of testing even in the absence of symptoms to detect asymptomatic infections (as informed by pilot evaluation). If a client accepts Xpert® testing, she will be instructed by the study nurse on how to self-collect a vaginal swab.
  Arms: Asymptomatic Only Testing; Universal Testing

SUMMARY:
The investigators will conduct a 3-arm individual-level RCT in Kisumu and Siaya, Kenya to compare perinatal outcomes associated with 3 models of STI testing and management in antenatal care. The investigators will enroll 3132 pregnant women and randomize 1:1:1 to receive standard-of-care (syndromic management only without CT, NG, or TV testing) vs. CT, NG, and TV testing using Xpert® assays universally vs. only among women without STI symptoms. All women with STIs detected and/or symptoms per Ministry of Health algorithms will receive immediate treatment, EPT per national guidelines, and tests of cure. All participants will be enrolled during routine antenatal care and followed through 9-months postpartum. The investigators will quantify and compare a composite outcome of pregnancy loss/stillbirth, PTB, LBW, SGA, and neonatal death, between randomization arms, in addition to several secondary and exploratory outcomes.

DETAILED DESCRIPTION:
In Aim 1, the investigators will conduct a 3-arm individual-level RCT in Kisumu and Siaya, Kenya to compare perinatal outcomes associated with 3 models of STI testing and management in antenatal care. The investigators will enroll 3132 pregnant women and randomize 1:1:1 to receive SOC (syndromic management only without CT, NG, or TV testing) vs. CT, NG, and TV testing using Xpert® assays universally vs. only among women without STI symptoms. All women with STIs detected and/or symptoms per Ministry of Health algorithms will receive immediate treatment, EPT, and tests of cure per national guidelines. All participants will be enrolled during routine antenatal care and followed through 9-months postpartum. The investigators will quantify and compare a composite outcome of pregnancy loss/stillbirth, PTB, LBW, SGA, and neonatal death, between randomization arms, in addition to several secondary and exploratory outcomes.

Antenatal clinic selection for RCT (Aim 1): The investigators conducted a landscape analysis of antenatal clinics in Kisumu and Siaya, Kenya as part of our team's ongoing PrEP studies. The investigators gathered data on the clients who attend antenatal care (e.g., HIV prevalence), the types of STI/HIV services offered (e.g., dual HIV and syphilis testing), and availability of the GeneXpert® platform. The investigators selected 9 high-volume clinics (>350 antenatal clients annually); all clinics must provide syndromic STI management per national guidelines, have a laboratory that runs Xpert® assays, and provide a full range of antenatal services (e.g., syphilis and HIV testing). The investigators consulted with county health officials, facility in-charges, and laboratory staff, who have assured us that providing Xpert® STI testing on existing GeneXpert® machines in facilities is possible (see letters of support from County Health Directors).

Study population and eligibility criteria (Aim 1): 3132 pregnant women seeking antenatal care will be recruited from 9 routine ANC facilities in Kisumu and Siaya, Kenya, to participate in the randomized trial. Eligibility criteria include identifying as a cisgender woman, seeking antenatal care that day, planning to receive antenatal and postnatal care at that clinic, and being willing and able to provide informed consent. The investigators will not exclude clients who report intimate partner violence from enrolling in the study as they may especially benefit from STI services.76. The investigators will also not exclude women based on age, HIV status, or gestational age at enrollment to produce findings based on a study sample most representative of the underlying population of antenatal clients in the region as these data will be most useful for policy decisions.

Recruitment, screening and enrollment of antenatal clients (Aim 1): At each clinic, enrollment will occur over a 14-month period (~25 antenatal clients enrolled per month, with seasonal variability) with an approximately 12-month follow-up period. Following registration at the clinic, study nurses will recruit clients and determine eligibility. Based on our recent studies in antenatal clinics in/near Kisumu, median gestational for clients seeking antenatal care is 24 weeks which is later than inclusion criteria of ongoing studies using Xpert® testing in other settings. Following screening consent, a brief form will capture age, HIV status, eligibility characteristics, and willingness to consent to join the study. Following written informed consent for participation, clients will be enrolled and assessed for demographic and behavioral characteristics, sexual history, education, marital status, income, relationship characteristics, HIV status, and clinical characteristics (e.g. pregnancy history, etc). Recruitment strategies will include collaborating with clinic staff and enrolled participants who will refer other clients who meet eligibility criteria. Recruitment materials will educate antenatal clients about STI risk based on available data, risks of having a partner of unknown STI status, and will emphasize the benefits of STI screening.

Randomization procedures (Aim 1): Randomization will occur following all routine antenatal procedures and enrollment into the study. Block randomization (1:1:1) in random sized blocks of no more than 9, stratified by recruitment site and HIV status at enrollment to ensure balance of arms within sites, will be overseen by the study biostatistician. Study nurses will be given randomly generated treatment allocations (SOC or universal testing or only asymptomatic testing) within sealed opaque envelopes. Once a participant has consented to enter the trial, an envelope will be opened, and the participant will be assigned the treatment allocation. The randomization code will be maintained by the Study Coordinator at the study site. Once assigned, the randomization allocation will be unblinded. To minimize the influence of the unblinded nature of the study on outcomes, ongoing data monitoring will not include information about endpoints disaggregated by site or arm. Only the study statistician will review data on study endpoints by arm or site.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as a cisgender woman
* Seeking antenatal services from the clinic
* Planning to receive antenatal and postnatal care at the clinic
* Willingness to receive syndromic STI screening and HIV/syphilis testing per national guidelines
* Able and willing to provide informed consent for participation

Exclusion Criteria:

* Male gender
* Not seeking antenatal services from the clinic
* Not planning to receive antenatal and postnatal care at the clinic
* Not willing to receive syndromic STI screening and HIV/syphilis testing per national guidelines
* Not able or willing to provide informed consent for participation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 3132 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Perinatal outcomes | 6 weeks postpartum
  Binary endpoint (Yes/No) of a composite of fetal loss, PTB<37 weeks gestation, SGA <10th percentile, and neonatal death compared between randomization arms

SECONDARY OUTCOMES:
EPT outcomes and factors | At each follow up visit
  Binary endpoint (Yes/No) of whether participant offered EPT to partner and if partner took EPT medications in intervention arm only
Quality of Care | At each follow-up visit
  Binary endpoints (Yes/No) based on MEASURE Evaluation's indicators for QOC in reproductive health (eg Did provider ask if you were having a problem with your FP method?) compared between randomization arms
CT/NG/TV prevalence and cofactors | 6 weeks postpartum
  Frequency of CT/NG/TV detection (Yes/No) at 6-weeks postpartum compared between randomization arms
Maternal HIV incidence | 9 months postpartum
  Frequency of HIV diagnosis at follow-up visits compared between randomization arms
Vertical HIV transmission | 9 months postpartum
  Frequency of HIV diagnosis among infants born to WLHIV at follow-up visits compared between randomization arms
Individual perinatal outcomes | 6 weeks postpartum
  Binary endpoint (Yes/No) of fetal loss, PTB<37 weeks gestation, SGA <10th percentile, and neonatal death, separately, compared between randomization arms
Antimicrobial resistence | 9 months postpartum
  Binary endpoints (Yes/No) of NG antimicrobial resistance detected among any NG infections

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Pintye, RN, MPH, PHD, Principal Investigator — University of Washington
Locations (8):
- Kenya (8):
  - Homa Bay Teaching and Referral Hospital, Homa Bay
  - Rachuonyo South Sub County Hospital, Homa Bay
  - Rangwe Sub County Hospital, Homa Bay
  - Chulaimbo County hospital, Kisumu
  - Kisumu County Hospital, Kisumu
  - Lumumba Sub County hospital, Kisumu
  - Migosi Sub County Hospital, Kisumu
  - Yala sub County Hospital, Yala

IPD SHARING:
Plan to Share IPD: No